CLINICAL TRIAL: NCT02963779
Title: A 2-Part, Safety, Tolerability, and Pharmacokinetic Study of LY2775240 in Healthy Subjects
Brief Title: A Study of LY2775240 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 16450; I8W-MC-PDBA (Other: Eli Lilly and Company)
Record Dates: First submitted 2016-11-10; First posted 2016-11-15 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Healthy
MeSH Terms: interventions — apremilast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- LY2775240 (Part A) (Experimental): Escalating oral doses of LY2775240 administered in healthy participants
  Interventions: Drug: LY2775240
- LY2775240 (Part B) (Experimental): Oral dose of LY2775240 in healthy participants
  Interventions: Drug: LY2775240
- Placebo (Part A) (Placebo Comparator): Placebo administered orally in healthy participants
  Interventions: Drug: Placebo
- Apremilast (Part B) (Active Comparator): Oral dose of apremilast in healthy participants
  Interventions: Drug: Apremilast

INTERVENTIONS:
Drug: LY2775240 — Administered orally
  Arms: LY2775240 (Part A); LY2775240 (Part B)
Drug: Placebo — Administered orally
  Arms: Placebo (Part A)
Drug: Apremilast — Administered orally
  Arms: Apremilast (Part B)

SUMMARY:
This study is conducted to determine the side effects related to LY2775240 given orally to healthy participants. Blood tests will be done to check how much LY2775240 is absorbed into the bloodstream and how long the body takes to get rid of it. Each participant will enroll in either Part A or Part B of the study, which will last about 14 weeks and 8 weeks respectively, including screening.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy adult male or a female who cannot get pregnant
* Have a screening body mass index (BMI) of greater than 18 and less than or equal to 32 kilograms per meter square (kg/m²), inclusive
* Have normal blood pressure, pulse rate, electrocardiogram (ECG) and medical test results that are acceptable for the study

Exclusion Criteria:

* Are currently participating in or completed a clinical trial within the last 30 days from a clinical trial or any other type of medical research judged to be incompatible with this study
* Have known allergies to compounds or drugs similar to LY2775240 or apremilast
* Have previously participated or withdrawn from this study
* Have or used to have health problems or medical test results or ECG readings that, in the opinion of the doctor, could make it unsafe to participate, or could interfere with understanding the results of the study

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-12; Primary Completion 2017-10-05 (Actual); Study Completion 2017-10-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline through to final follow-up at approximately Week 14

SECONDARY OUTCOMES:
Pharmacokinetics: Area Under the Concentration Curve (AUC) of LY2775240 | Baseline through Day 5
Pharmacokinetics: Time to Maximal Blood Concentration of LY2775240 | Baseline through Day 5
Pharmacokinetics: Maximum Concentration of LY2775240 in Blood | Baseline through Day 5

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Singapore, Singapore